CLINICAL TRIAL: NCT02868216
Title: Management of Anger in Patients With ST Segment Elevation Acute Myocadial Infarction: A Randomized Clinical Trial
Brief Title: Management of Anger in Patients With Acute Myocardial Infarction (MAPAMI)
Acronym: MAPAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UP4985/14
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Results first posted 2019-11-05 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Anger Management Therapy

STUDY DESIGN:
Intervention Model Description: One group receives training for anger management, with guidance on infarction and physiology of anger and another group, does not receive.
Who Masked: Outcomes Assessor
Masking Description: Blinding occurs only in relation to the evaluator of endothelial function
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anger management training (Experimental): treatment group- Two monthly sessions will address the events triggering anger, the physiology of anger and the influence on the cardiovascular system, the dimesions of anger: cognitive, emotional and behavioral.
  Interventions: Behavioral: anger management training
- Without management training (No Intervention): No anger management training

INTERVENTIONS:
Behavioral: anger management training
  Arms: anger management training

SUMMARY:
Stress, anger and depressed can operate as a trigger to an Acute Coronary Syndrome. It is often found in the literature that patients refer excessive anger, anxiety, sadness, pain or acute stress before the acute myocardial infarction (AMI). Moreover, a recent meta-analysis reported a strong association between the occurrence of AMI and many of these acute emotions.

Anger is a common manifestation of psychological stress and could trigger off an atherogenic process through several mechanisms.

Coronary atherosclerosis features narrowing of coronary arteries on account of endothelial thickening caused by the build up of atheromatous plaques. It is a process characterized by inflammatory and fibroproliferative response of the artery wall, caused by continuous aggression to its surface and whose thickening, evoked by the evolution of fat streaks atherosclerotic lesions, until fiber plaques is quite slow. Endothelial dysfunction also results in the loss of natural anti-thrombotic properties involved in the endothelium patency.

According to a study performed by our group, anger management was significantly lower among patients with CAD when compared to those without CAD, and the occurrence of major cardiovascular events (MACE) was significantly higher in patients presented with lower anger control. Both associations were independent from traditional risk factors, occurrence of previous events or another anger aspects. Thus, this study was designed in order to evaluate the effect of the "cognitive training to anger management " on endothelium-dependent vasodilation of the arm artery in patients with acute myocardial infarction with ST segment elevation submitted to primary coronary intervention.

DETAILED DESCRIPTION:
ANGER EVALUATION:

Anger will be assessed by the Spielberger State-Trait Anger Expression Inventory (STAXI). This instrument was developed to evaluate the expression of anger components and their role in a variety of medical conditions. These are statements to be assessed on a Likert scale of 4 points. Individuals are asked about the intensity of his anger, and how often experience this emotion.

The anger trait measures individual differences in willingness to experience anger. It is evaluated through 10 questions, with their scores between 10 and 40 points. It is divided in temperament and anger reaction. Anger expression provides a general index on the frequency with which anger is experienced, expressed, suppressed or controlled and is evaluated with three subscales: anger inside, when angry feelings are repressed or stored; anger-out, when the individual expresses anger toward other persons or objects in the environment; and anger management (control) which measures the frequency with which each individual tries to control the expression of raiva. Each of these subscales is assessed by eight questions, ranging from 32 to 64 points. The total score for the expression of anger is evaluated by the results: Total + in total off - control +16.

Randomization All patients were evaluated during hospitalization for AMI, but only those anger control score were less than 27 points were invited to participate. A randomization list was obtained by random.org site and were generated sequential envelopes, sealed and numbered which were opened in order day in assessment of endothelial function.

Endothelial function Endothelial dysfunction is an early dysfunctional vascular responses observed in tissue prone to develop atherosclerosis and is also associated with vessel with atherosclerosis in later stages. The evaluation of endothelial function will be performed by researchers "blinded" as to treatment group. The endothelium-dependent vasodilation of the brachial artery will be evaluated by ultrasound with a linear transducer 3-12 MHz (EnVisor CHD, Philips, Bothell, WA, USA), being held automated measurements of vessel diameter to own the equipment used software. The evaluations will be conducted in the mornings after fasting for 12 hours under controlled temperature (22 ° C). After ten minutes of images of the brachial artery rest will be recorded with the linear transducer placed above the antecubital fossa continuously for one minute (basal). The sphygmomanometer is placed on the arm and inflated up to 50 mmHg limit above systolic blood pressure for five minutes, and the change in diameter of the brachial artery after 60 seconds of cuff deflation will be compared with the basal diameter. The images of the vessel diameter at end-diastole (identified by R wave of the ECG) will be digitized and recorded at intervals of 3 seconds throughout the procedure, and subsequently analyzed off-line using software itself equipamento41.

ANGER TREATMENT:

session 1 -Participants are asked what usually makes them angry. The "triggers" of anger are identified; the relationship between rabies and cardiovascular physiology is explained. According to Lipp and Malagris19 (p.115), "anger changes the way the body works, changes breathing, pressure increases, etc. When a person feels anger, the physical reaction that occurs is automatic and unplanned, it is difficult control, but the identification of triggers before the emotion sets in, will help to prevent it. Identifying and understanding anger in three dimensions: cognitive, emotional, and behavioral Think before acting Behavior is the final step, which you do not need be damaging.

Session 2 - Participants are reminded of "elicitor rabies events". Investigate the situations that felt anger during the month and what they thought. To point out how the cognitions, that is, how one interprets the facts of life leads to different emotions. How anger behavior is directly linked to the interpretations people give to events; It is important to improve the way you evaluate events and the world around you. Closing: Deep Breathing Exercise Technical Time-Out: isolate yourself from the situation that generates anger to take control.

The control group patients will not receive any anger managementtraining.

STATISTICAL ANALYSIS

The minimum sample size was calculated in 88 patients to detect a 1% difference in flow-mediated dilation between the two study groups, with an average standard deviation of 1.67%, p <0.05 and statistical power of 90 %. The data are presented as means and confidence intervals (95% CIs), unless otherwise specified. All analyzes will be based on the principle of intention to treat, and will be conducted by researchers who do and whether or not the cognitive training for control of anger. Repeated measures of analysis of variance will be performed to determine differences in flow-mediated dilation (primary endpoint) and all secondary outcomes between the two groups over time, using a conservative F test for the interaction between time and study group ( SPSS software, version 18).

The Geisser correction for the F test is used to adjust the degrees of freedom for the roundness deviation (one of the conditions of the repeated measures analysis of variance [ANOVA]). logarithmic transformation of the data will be undertaken as appropriate. Fisher's post hoc analysis for unpaired and paired data will be performed and interpreted using the Bonferroni-Holm adjustment for multiple comparisons.

The post correlation hoc analysis (by the Spearman rank-correlation method) will be performed to evaluate the relationship between the change in flow-mediated dilation of the baseline to 3 months and the changes in the anger control scores assessed by STAXI from the beginning up to 3 months. Differences between categorical variables are calculated using the chi-square test. A value of P-tailed <0.05 is considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

acute st elevation myocardial infarction

Exclusion Criteria:

* dementia, cognitive dysfunction,
* bypass surgery previous or during the study periods living from more 200 Km from hospital

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Moura Schmidt, PhD, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmidt KES, de Quadros AS, Eibel B, Aires AM, Gottschall CAM, Moura MRS, Schmidt MM. The Influence of Cognitive Behavioral Intervention for Anger Management on Endothelial Function in Patients With Recent Myocardial Infarction: A Randomized Clinical Trial. Psychosom Med. 2022 Feb-Mar 01;84(2):224-230. doi: 10.1097/PSY.0000000000001039. PMID 34840289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: dates of the recruitment: 09/15/2015 to 07/15/2017 patients with AMY in this period: 707
Pre-assignment Details: Patients submitted to myocardial revascularization surgery, with acute or chronic infections, need for mechanical ventilation or other complications were excluded; those with delirium, cognitive or mental difficulties, aged ≥ 80 years; and also, unable to comply with follow-up visits or who refused to participate.
Groups:
- Anger Management Training: treatment group- Two monthly sessions will address the events triggering anger, the physiology of anger and the influence on the cardiovascular system, the dimesions of anger: cognitive, emotional and behavioral.
  anger management training
Period: Overall Study
Arm/Group | Anger Management Training | Without Management Training
Started | 43 | 47
Completed | 35 | 41
Not Completed | 8 | 6
Not completed — Death | 0 | 1
Not completed — coronary artery bypass | 1 | 0
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anger Management Training | Without Management Training | Total
Number analyzed (Participants) | 35 | 41 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (9) | 58 (10) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 27 | 32 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 29 | 36 | 65
  Race: Afro-descendant | 6 | 5 | 11
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 35 | 41 | 76

OUTCOME MEASURES:

1. Primary Outcome: Difference in Flow-mediated Dilation in the Brachial Artery in the Base and After the Treatment.
Description: Inter group difference in flow-mediated dilation in the brachial artery in the baseline and after the treatment (about Three months after the first).
  Vasodilatation of the endothelium-dependent brachial artery was evaluated by ultrasound using a 3-12 MHz linear transducer. Three images of the basal diameter (BD) of the brachial artery at the end of the diastole were acquired, as well as the mean velocity of the baseline arterial flow, with the linear transducer positioned 5 cm above the antecubital fossa. Subsequently, the sphygmomanometer was placed in the arm and inflated 50 mmHg above baseline systolic blood pressure for five minutes. After that, 3 images of the arterial diameter were acquired up to 80 seconds of the deflation of the cuff (post-occlusion diameter- PD), as well as the average of the arterial flow velocity. Flow-dependent vasodilation responses were expressed as a percentage variation from the baseline brachial diameter (PD-BD/ BD x 100).
Time Frame: three months after the first evaluation
Population: means and standard deviations after treatment
Measure: Mean (Standard Deviation); unit: percent change dilatation
Arm/Group | Anger Management Training | Without Management Training
Number analyzed (Participants) | 35 | 41
percent change dilatation | 11.24 (5.10) | 7.70 (4.40)
Statistical Analysis 1: Comparison: Anger Management Training vs Without Management Training; Test type: Other; p = 0.05, ANOVA; Mean Difference (Final Values) = 2.30, 95% CI 2-sided [0.63 to 3.98], Standard Deviation 0.84

ADVERSE EVENTS:
Groups:
- Intervention: Major adverse cardiovascular events: totally of death, myocardial infarction, percutaneous coronary intervention in intervention group
- Controls: Major adverse cardiovascular events: totally of death, myocardial infarction, percutaneous coronary intervention in control group
Arm/Group | Intervention | Controls
All-Cause Mortality (participants affected / at risk) | 2/33 | 1/39
Serious Adverse Events (participants affected / at risk) | 5/33 | 2/39
Other Adverse Events (participants affected / at risk) | 2/33 | 1/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=33) | Controls (N=39)
Major adverse Cardiovascular events (Cardiac disorders) | 5 | 2 — Mortality, myocardial infarction and percutaneous coronary intervention
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=33) | Controls (N=39)
Percutaneous coronary intervention (Cardiac disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes